CLINICAL TRIAL: NCT06632964
Title: An Open-label, Single-arm Exploratory Clinical Trial Aimed At Assessing the Efficacy and Safety of VT-101 for the Treatment of Non-muscle Invasive Bladder Cancer
Brief Title: A Clinical Trial Aimed At Assessing the Efficacy and Safety of VT-101 for the Treatment of Non-muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2024-KL364-02
Record Dates: First submitted 2024-09-27; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-08

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: Oncolytic virus; Non-muscle invasive bladder cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VT-101 (Experimental): The registered patients will receive oncolytic adenovirus VT-101 therapy for the non-muscle invasive bladder cancer by intravesical instillation.
  Interventions: Biological: Recombinant oncolytic adenovirus injection solution of VT-101

INTERVENTIONS:
Biological: Recombinant oncolytic adenovirus injection solution of VT-101 — Active ingredient: VT-101 recombinant oncolytic adenovirus Specifications: 2×10^10 IFU/ml, 0.5ml/ capsule Method of administration: intravesical perfusion

SUMMARY:
This is an experimental study to evaluate the efficacy and safety of VT-101 for the treatment of non-muscle invasive bladder cancer

DETAILED DESCRIPTION:
The investigators designed a clinical study and divided the trial into two phases.

Phase 1(climbing test): The first dose group (2×10^10 IFU) in the ramp-up phase is the accelerated titration dose group, which will include one patient. During the observation period of dose-limiting toxicity (DLT) in the accelerated titration phase (set as 7 days after initial drug administration for each participant), if a grade 2 or higher treatment-related adverse event (TRAE) is observed, or when escalating to the second dose group (5×10^10 IFU dose group), it will transition to a conventional escalation phase using a 3+3 dose escalation design: If no DLT occurs in 0/3 participants during the observation period, it will escalate to the next dose; if DLT occurs in 1/3 participants during the observation period, an additional three participants will be enrolled at this dosage level simultaneously. If no DLT occurs among these additional three participants during their observation period (total of 1/6 subjects with DLT), it will proceed to the next dose group. If ≥2/6 participants experience DLT, then the ramp-up trial will terminate and a lower dosage level below current level will be selected for dosing expansion stage. Alternatively, based on existing clinical data, the investigators may redefine ramp-up doses. If no DLT occurs in 0/3 or 1/6 of participants during the observation period of the 10×10^10 IFU dose group, the investigators determine whether to continue increasing ramp-up doses and ultimately determine dosages for expansion stage based on exploration results from ramp-up phase. Participants who do not experience DLT during ramp-up phase can continue receiving study drug at same dosage via intravesical instillation once weekly for six consecutive weeks (including initial administration). Subsequent administration is determined by the investigators monthly and should not exceed one year unless disease progression or recurrence occurs, intolerable toxicity develops, participant withdraws informed consent or dies, the investigator deems continued treatment inappropriate or other termination criteria are met according to earliest.

Phase 2:During the expansion phase, approximately 8-10 participant will be enrolled based on the recommended dose from the escalation phase. The number of participant may be adjusted by the investigators based on existing trial data, and non-resectable high-risk and very high-risk NMIBC patients may also be included in the expansion phase study. The dosing plan for the expansion phase is as follows: multiple administrations once a week through intravesical instillation for six consecutive weeks. Subsequent administration frequency will be determined by the investigators (once a month, up to a maximum of one year) or until disease progression or recurrence occurs, intolerable toxicity arises, participant withdraws informed consent or dies, the investigator deems it inappropriate to continue treatment, or other termination criteria are met with priority given to events occurring first.

Dose-Limiting Toxicity (DLT) is defined as an event related to the investigational drug that meets any of the following criteria during the observation period:

1. Any toxicity ≥ Grade 3 except for fatigue lasting ≤3 days or fatigue and weakness that can be relieved through rest or self-adjustment; clinically insignificant reversible laboratory abnormalities ≥ Grade 3.
2. Any toxicity that cannot recover to ≤ Grade 1 baseline level within seven days after discontinuation of dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including 18 and 75 years old), male or female;
2. Patients with non-muscle-invasive bladder cancer (NMIBC) confirmed by histopathological examination results (pathological stage: high-grade Ta or any T1 level papillary carcinoma or cystoscopic random biopsy confirmed presence of bladder in situ carcinoma (CIS) (with or without papillary carcinoma): according to the results of the biopsy taken within 8 weeks before the first treatment according to the study. If multiple bladder biopsies are needed to confirm eligibility, the last biopsy must be taken within 8 weeks.

   For patients with high-risk disease at the second TURBT, defined as high-grade Ta/T1 lesions, the subject must completely remove all visible tumors before enrollment and be recorded at the baseline cystoscopy.

   The results of the cellular pathology examination for high-grade urothelial carcinoma must be negative before enrollment, excluding those with unresectable high-risk and extremely high-risk NMIBC in the dose-escalation stage.

   CIS does not require complete removal, but must be completely removed along with papillary carcinoma before enrollment, and be recorded at the baseline cystoscopy. No requirement is made for negative urine cytology results for malignant cells.

   For those with unresectable high-risk and extremely high-risk NMIBC included in the dose-escalation stage, urine cytology results for malignant cells may not be required to be negative before enrollment.

   When the investigator assesses the subject as medically unfit for TURBT or radical cystectomy or the subject refuses TURBT or radical cystectomy after consulting a urologist, the subject may also participate in this study.
3. Moderate, high risk and very high risk NMIBC; Specific definitions are as follows:

   1. Medium-risk NMIBC:

      ● Does not meet the conditions of low risk, high risk, and very high risk groups, and does not have CIS
   2. High-risk NMIBC:

      * T1 HG/G3 tumors without CIS and not eligible for the very high risk group
      * Tumors present CIS and do not meet the conditions of the very high risk group
      * Ta LG/G2 or TI G1, no CIS, and three clinically relevant risk factors Ta HG/G3 or TI LG, without CIS, and with at least two clinically relevant risk causes plain
      * TI G2, without CIS and containing at least one clinically relevant risk factor c.very high risk NMIBC:
      * Ta HG/G3 with CIS and three clinically relevant risk factors ●TI G2 with CIS and at least two clinically relevant risk factors
      * TIHG/G3, CIS, with at least one clinically relevant risk factor ●TIHG/G3, CIS, with three clinically relevant risk factors
      * CIS in the prostatic urethra
      * Urothelial carcinoma with undesirable histological variation subtype
      * Accompanied by vascular lymphatic invasion

      Note: Clinically relevant risk factors include:
      1. Age≥ 70 years old;
      2. Multiple papillary tumors;
      3. Diameter≥ 3cm. Subtypes of adverse histological variation include: urothelial carcinoma with partial squamous or adenoid or trophoblastic differentiation, micropapillary urothelial carcinoma, nested nested nested variant (including large nested variant), and microcystic variant urothelial carcinoma, plasmacytoid, giant cell, sigma-ring cell, diffuse, undivided Metastatic urothelial carcinoma, lymphoepitheliomatoid carcinoma, small cell carcinoma, sarcomatoid urothelial carcinoma, introneural secretory variant urothelial carcinoma.
4. The general status score of the American Eastern Oncology Consortium (ECOG) (Appendix 4) was 0 to 1;
5. Expected survival≥ 2 years;
6. The subjects have adequate organ and bone marrow function, meeting the following laboratory test criteria (Note: If an individual laboratory test result does not meet the criteria, a repeat screening is allowed):

   Complete blood count: absolute neutrophil count (ANC) ≥ 1.5×109/L, white blood cell count (WBC) ≥3.0×109/L, platelet count (PLT) ≥75×109/L, hemoglobin (Hb) ≥90g/L (Note: No blood components, cell growth factors, etc. may be used for interventional treatment within 14 days prior to the test to ensure that the test results meet the above requirements).

   Liver function: Serum total bilirubin (TBIL) ≤ 1.5 x ULN, albumin (ALB) ≥30 g/L; No liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN; Liver metastasis, ALT and AST need ≤5.0 x ULN; Kidney function: Serum creatinine (Scr) ≤ 1.5 x ULN, or creatinine clearance rate ≥ 50 mL/min (creatinine≥ 1.5 x ULN, creatinine clearance rate will be calculated according to Cockcroft-Gault formula.); Coagulation function: International normalized ratio (INR) ≤1.5 x ULN or prothrombin time (PT) ≤ 1.5 x ULN, and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
7. The results of blood pregnancy test performed by women of childbearing age within 7 days before treatment were negative. Female participants of reproductive age, as well as male participants whose partners are women of reproductive age, must agree to use at least one medically approved contraceptive method (such as surgical sterilization, oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicide) for the entire study period and for at least 6 months after the last study drug treatment. Fertile women in this program are defined as sexually mature women who have not undergone hysterectomy or bilateral oophorectomy; or spontaneous menopause that has not lasted 24 months (amenorrhea after cancer treatment does not exclude fertility), that is, menstruation at any time in the 24 consecutive months prior to screening);
8. Male subjects must agree not to donate sperm during treatment and for at least 6 months after the last treatment;
9. The subjects fully understand and know the whole study process, voluntarily participate in the study, sign the informed consent, and the expected compliance is good.
10. During the study period, patients must be willing to comply with the study requirements for cystoscopy, urine cytology, urography, biopsy (TURBT or other excision for all Ta/T1 diseases). For these procedures, patients who withdraw their consent will withdraw from the trial.

Exclusion Criteria:

1. A current or past history of muscular invasive (T2 or higher stage) or locally advanced (T3/T4, any N) or metastatic bladder cancer;
2. Urothelial carcinoma of the upper urogenital tract (kidney, renal collecting system, ureter) or prostatic urethra (including urethral CIS) in the 24 months prior to enrollment;
3. Cystoscopy orimaging examination confirmed the current bladder perforation;
4. Prior systemic treatment, radiation therapy, or surgery for bladder cancer during screening, in addition to TURBT or bladder biopsy. Intravesical perfusion within 8 weeks prior to initiation of study therapy, with the exception of a single infusion of cytotoxic drugs (e.g. mitomycin C, gemcitabine, pirarubicin, and epirubicin) immediately after TURBT surgery;
5. Past treatment with oncolytic virus drugs or similar drugs;
6. Concurrent severe medical conditions, including but not limited to severe heart disease, cerebrovascular disease, uncontrolled diabetes, severe infection, active digestive ulcer, or uncontrolled high blood pressure (defined as systolic/diastolic blood pressure ≥150/100 mmHg after treatment with standardized antihypertensive drugs, or one of them); Angina pectoris in the last 3 months; Myocardial infarction or cardiac insufficiency within 1 year prior to enrollment (NYHA rating: Heart function ≥II, see Appendix 2); Severe arrhythmias requiring medical treatment; Left ventricular ejection fraction (LVEF) ≤ 50%; Adjusted for QTc interval (Fridericia formula) ≥ 480 ms, or risk factors present at the tip of torsified ventricular tachycardia, such as clinically significant hypokalemia as determined by the investigator, family history of long QT syndrome, or family history of arrhythmia (such as preexcitation complex);
7. Patients who are expected to have major surgery during the study period (including the screening period);
8. The subject has an active infection or unexplained fever≥ 38.5 ℃ during screening or before the first dose;
9. Subject with congenital or acquired immune deficiency (such as HIV infection), syphilis antibody positive or active hepatitis B: Hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb] positive with ≥ 1000 copies of HBV-DNA [cps]/mL or higher than the upper limit of normal detection; Or test positive for hepatitis C antibodies, and HCV-RNA is higher than the upper limit of normal test values;
10. Had received any of the following treatments within a specified time frame prior to enrollment: a. Had undergone major surgery (whether or not related to the tumor) within 4 weeks, except for minimally invasive surgery under gastroenteroscopy; b. Within 4 weeks Extended radiotherapy, or local radiotherapy within 2 weeks (investigators can determine the appropriate enrollment time based on the recovery of toxicity after radiotherapy); c. Participating in other therapeutic/interventional clinical trials within 4 weeks or currently; d. Received any local or systemic anti-tumor therapy (including anti-tumor Chinese medicines and Chinese adult drugs) within 4 weeks or within 5 half-lives of the drug (calculated as a shorter time);
11. Presence of toxicity from prior antitumor therapy that has not returned to CTCAE 5.0 level 0 or 1 or levels specified in the inclusion or exclusion criteria prior to initial administration (excluding alopecia, skin pigmentation, and non-clinically significant and asymptomatic laboratory abnormalities);
12. Received immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc., within 2 weeks before the first dose;
13. Allergic to adenovirus or any component of the test drug;
14. The subject has a known history of psychotropic substance abuse, alcohol abuse, or drug use;
15. History of other malignancies within the last 5 years, except cured basal cell carcinoma of the skin, cured cervical carcinoma in situ, and cured thyroid carcinoma in situ;
16. Subjects with an active autoimmune disease or a history of an autoimmune disease that may recur, but subjects with the following conditions are admitted:

    1. Patients with type 1 diabetes whose condition is stable after treatment with stable doses of insulin;
    2. hypothyroidism (if controlled with hormone replacement therapy alone);
    3. controlled and stable celiac disease;
    4. Skin diseases that do not require systemic treatment (e.g. vitiligo, psoriasis, alopecia);
    5. any other disease that will not recur in the absence of an external trigger.
17. Patients need to use corticosteroids (prednisone≥ 10 mg/ day or equivalent dose of the same drug) or any other condition requiring systemic immunosuppressant treatment for 4 weeks prior to initial dosing. However, participants who are currently or have previously used the following steroid regimens may be enrolled:

    1. adrenal substitute steroid (prednisone ≤10 mg/ day or equivalent dose of similar drugs);
    2. Systemic absorption of very small amounts of local, ocular, intra-articular, intranasal or inhaled corticoid solid alcohol.
18. Pregnant or lactating women, or male and female subjects who planned to have children during the trial period (from screening visit to 6 months after the last dosing). Any pregnancy that occurred during the test Participants need to withdraw from the study;
19. Persons who need to receive live vaccine within 30 days before the first dose and during the expected study period;
20. The investigator considers that the subjects have other factors that make them unfit to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of possible adverse events after intravesical instillation of VT-101 | 3 months after VT-101 intravesical instillation
  To evaluate the safety of VT-101 in the treatment of non-muscular invasive bladder cancer.Changes in vital signs, physical examination results, ECOG performance score, laboratory tests, and 12-lead electrocardiogram before, after, and during treatment.
The proportion of patients who suspend or discontinue treatment due to drug toxicity | 3 months after VT-101 intravesical instillation
  Dose-Limiting Toxicity (DLT) is defined as an event related to the investigational drug that meets any of the following criteria during the observation period:
  Any toxicity ≥ Grade 3 except for fatigue lasting ≤3 days or fatigue and weakness that can be relieved through rest or self-adjustment; clinically insignificant reversible laboratory abnormalities ≥ Grade 3.
  Any toxicity that cannot recover to ≤ Grade 1 baseline level within seven days after discontinuation of dosing.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | 3 months after VT-101 intravesical instillation
  To observe the efficacy of VT-101 after intravesical infusion.Complete Response (CR) is defined as either a) negative cystoscopy and negative urine cytology (including atypical) or b) negative cystoscopy, positive urine cytology and negative random bladder biopsy.
Partial Response (PR) Rate | 3 months after VT-101 intravesical instillation
  To observe the efficacy of VT-101 after intravesical infusion.Partial Response (PR) is defined as a reduction of the tumor by more than 50% over a period of not less than 4 weeks, which can be measured by either double-path or single-path measurements. (a) Double diameter measure1) Single lesion: tumor area (the product of the two largest vertical diameters of the mass) reduced by ≥50%; 2) Multiple lesions: the sum of the product of the two largest vertical diameters of multiple masses is reduced by more than 50%. (b) Single diameter measurement: The measured value of linear mass is reduced by more than 50%.
Stable Disease (SD) | 3 months after VT-101 intravesical instillation
  To observe the efficacy of VT-101 after intravesical infusion.Stable disease (SD) is defined as being somewhere between partial remission and disease progression.
Progressive Disease (PD) | 3 months after VT-101 intravesical instillation
  To observe the efficacy of VT-101 after intravesical infusion.Progressive Disease (PD) is defined as a 20% increase in the sum of the longest tumor diameters or the appearance of one or more new lesions compared to the sum of the smallest tumor longest diameters recorded after the start of treatment.
Disease-Free Survival (DFS) | 3 months after VT-101 intravesical instillation
  To observe the efficacy of VT-101 after intravesical infusion.Disease-free survival (DFS) was defined as continuous CIS≥6 months from the time of first dosing to the onset of any Ta, any T1 grade, new CIS, disease progression, cystectomy, change in treatment due to disease deterioration, or death (any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Junnian Zheng, M.D/Ph.D, Study Director — The Affiliated Hospital of Xuzhou Medical University; Hailong Li, M.D/Ph.D, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Meng Lu, Ph.D, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaurasiya S, Fong Y, Warner SG. Oncolytic Virotherapy for Cancer: Clinical Experience. Biomedicines. 2021 Apr 13;9(4):419. doi: 10.3390/biomedicines9040419. PMID 33924556
- [Background] Packiam VT, Lamm DL, Barocas DA, Trainer A, Fand B, Davis RL 3rd, Clark W, Kroeger M, Dumbadze I, Chamie K, Kader AK, Curran D, Gutheil J, Kuan A, Yeung AW, Steinberg GD. An open label, single-arm, phase II multicenter study of the safety and efficacy of CG0070 oncolytic vector regimen in patients with BCG-unresponsive non-muscle-invasive bladder cancer: Interim results. Urol Oncol. 2018 Oct;36(10):440-447. doi: 10.1016/j.urolonc.2017.07.005. Epub 2017 Jul 26. PMID 28755959
- [Background] Burke JM, Lamm DL, Meng MV, Nemunaitis JJ, Stephenson JJ, Arseneau JC, Aimi J, Lerner S, Yeung AW, Kazarian T, Maslyar DJ, McKiernan JM. A first in human phase 1 study of CG0070, a GM-CSF expressing oncolytic adenovirus, for the treatment of nonmuscle invasive bladder cancer. J Urol. 2012 Dec;188(6):2391-7. doi: 10.1016/j.juro.2012.07.097. Epub 2012 Oct 22. PMID 23088985
- [Background] Chesney J, Puzanov I, Collichio F, Singh P, Milhem MM, Glaspy J, Hamid O, Ross M, Friedlander P, Garbe C, Logan TF, Hauschild A, Lebbe C, Chen L, Kim JJ, Gansert J, Andtbacka RHI, Kaufman HL. Randomized, Open-Label Phase II Study Evaluating the Efficacy and Safety of Talimogene Laherparepvec in Combination With Ipilimumab Versus Ipilimumab Alone in Patients With Advanced, Unresectable Melanoma. J Clin Oncol. 2018 Jun 10;36(17):1658-1667. doi: 10.1200/JCO.2017.73.7379. Epub 2017 Oct 5. PMID 28981385
- [Background] Ribas A, Dummer R, Puzanov I, VanderWalde A, Andtbacka RHI, Michielin O, Olszanski AJ, Malvehy J, Cebon J, Fernandez E, Kirkwood JM, Gajewski TF, Chen L, Gorski KS, Anderson AA, Diede SJ, Lassman ME, Gansert J, Hodi FS, Long GV. Oncolytic Virotherapy Promotes Intratumoral T Cell Infiltration and Improves Anti-PD-1 Immunotherapy. Cell. 2017 Sep 7;170(6):1109-1119.e10. doi: 10.1016/j.cell.2017.08.027. PMID 28886381
- [Background] Andtbacka RH, Kaufman HL, Collichio F, Amatruda T, Senzer N, Chesney J, Delman KA, Spitler LE, Puzanov I, Agarwala SS, Milhem M, Cranmer L, Curti B, Lewis K, Ross M, Guthrie T, Linette GP, Daniels GA, Harrington K, Middleton MR, Miller WH Jr, Zager JS, Ye Y, Yao B, Li A, Doleman S, VanderWalde A, Gansert J, Coffin RS. Talimogene Laherparepvec Improves Durable Response Rate in Patients With Advanced Melanoma. J Clin Oncol. 2015 Sep 1;33(25):2780-8. doi: 10.1200/JCO.2014.58.3377. Epub 2015 May 26. PMID 26014293
- [Background] Hamid O, Hoffner B, Gasal E, Hong J, Carvajal RD. Oncolytic immunotherapy: unlocking the potential of viruses to help target cancer. Cancer Immunol Immunother. 2017 Oct;66(10):1249-1264. doi: 10.1007/s00262-017-2025-8. Epub 2017 Jul 15. PMID 28712033
- [Background] Wei W, Zeng H, Zheng R, Zhang S, An L, Chen R, Wang S, Sun K, Matsuda T, Bray F, He J. Cancer registration in China and its role in cancer prevention and control. Lancet Oncol. 2020 Jul;21(7):e342-e349. doi: 10.1016/S1470-2045(20)30073-5. PMID 32615118
- [Background] Zheng R, Zhang S, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2016. J Natl Cancer Cent. 2022 Feb 27;2(1):1-9. doi: 10.1016/j.jncc.2022.02.002. eCollection 2022 Mar. PMID 39035212